CLINICAL TRIAL: NCT01515085
Title: MRI-Guided Laser-Induced Thermal Therapy for Cytoreduction of Inoperable Grade III/IV GLiomas Prior to Chemotherapy and Radiation
Brief Title: MRI-Guided Laser Induced Thermal Therapy
Acronym: LITT
Status: Terminated | Type: Observational
Why Stopped: PI elected to close study
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 0220110114
Record Dates: First submitted 2011-10-18; First posted 2012-01-23 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — Laser Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- biopsy proven glioma, no prior treatment
  Interventions: Procedure: laser interstitial thermal therapy

INTERVENTIONS:
Procedure: laser interstitial thermal therapy — residual gliomas either after debulking or biopsy evaluated for intervention with laser ablation prior to onset of adjuvant therapy
  Other Names: laser ablation; LITT

SUMMARY:
Does MR-guided laser interstitial thermal therapy (MRgLITT) prior to chemotherapy and/or radiation give patients a beneficial increase in overall survival? Laser induced thermal therapy (LITT) is a minimally invasive procedure for destroying tissue through generation of heat.

DETAILED DESCRIPTION:
Laser induced thermal therapy (LITT) is a procedure for destroying tissue through generation of heat. When used in conjunction with fiberoptic applicators, it offers an excellent means of minimally invasive surgery. As opposed to other thermal techniques like radio-frequency (RF) ablation, or cryo-ablation, LITT may be significantly faster and may exhibit sharper boundary of the thermal ablation zone. More importantly, LITT is highly compatible with MR imaging and when coupled with MR thermal imaging (MRTI) guidance, precise monitoring of the thermal ablation zone in order to avoid eloquent or critical structures is possible.

In this study, we propose to evaluate MR-thermal image guided laser interstitial therapy for the treatment of inoperable brain tumors as upfront therapy prior to initiation of chemotherapy and radiation. MR-thermal imaging (MRTI) will be used to provide information on thermal dose delivered to the target and be used to control laser delivery to prevent damage to critical structures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that have/will undergo MRgLITT for inoperable brain tumor.
* Tumor size < 3cm in transverse diameter for each planned applicator placement.
* Tumor size < 4 cm in largest dimension.
* Lesion(s) are clearly defined on pre-therapy contrast enhanced MRI scans as determined by the treating surgeon.
* Karnofsky Performance Scale score > 70.
* ECOG performance status of 2 or better.
* Biopsy proven histologic diagnosis of malignant glioma.

Exclusion Criteria:

* Patients with co-existing medical conditions with life expectancy < 1 year.
* Patients having received pre-ablation chemotherapy and/or radiation to lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain tumors receiving MR-guided laser ablation
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival | three years

SECONDARY OUTCOMES:
Overall survival | three years

CONTACTS AND LOCATIONS:
Overall Officials: Shabbar F Danish, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States